CLINICAL TRIAL: NCT01582321
Title: Investigation of the Influence of Gender on Cardiovascular Function and Inflammation
Brief Title: Investigation of the Influence of Gender on Cardiovascular Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11/LO/2038
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cardiovascular Function
Keywords: vascular ultrasound; flow cytometry; platelet aggregation
MeSH Terms: interventions — Typhoid-Paratyphoid Vaccines; Vi polysaccharide vaccine, typhoid; Cantharidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 Male (Experimental): 16 healthy male volunteers will be recruited. Primary and secondary outcome measures will be made on day 1, 3 and 4. At 24 and 72 hours prior to outcome measures on day 3 a cantharidin-soaked 1cm2 filter paper disc will be applied to participants forearm or back on leg for blister formation. Blister fluids will be harvested on day 3.
  Interventions: Drug: Cantharidin
- Part 1 Female (Experimental): 16 healthy female volunteers will be recruited. Primary and secondary outcome measures will be made on day 1, 3 and 4. At 24 and 72 hours prior to outcome measures on day 3 a cantharidin-soaked 1cm2 filter paper disc will be applied to participants forearm or back on leg for blister formation. Blister fluids will be harvested on day 3.
  Interventions: Drug: Cantharidin
- Part 2 Male (Experimental): 12 healthy male volunteers will be recruited. Primary and secondary outcome measures will be made on day 0, 1 and 2. At 8 hours prior to outcome measures on day 1 intra-muscular typhoid vaccine will be administered.
  Interventions: Biological: Typhoid vaccine
- Part 2 Female (Experimental): 12 healthy female volunteers will be recruited. Primary and secondary outcome measures will be made on day 0, 1 and 2. At 8 hours prior to outcome measures on day 1 intra-muscular typhoid vaccine will be administered.
  Interventions: Biological: Typhoid vaccine

INTERVENTIONS:
Biological: Typhoid vaccine — The typhoid vaccine is composed of purified polysaccharide from S. typhi capsule 25 micrograms contained in 0.5 ml solution
  Other Names: Typhim Vi®
  Arms: Part 2 Female; Part 2 Male
Drug: Cantharidin — 0.1% cantharidin solution in acetone from 0.7% stock solution of cantharone is prepared and applied immediately. 10 μl of cantharidin per disc.
  Other Names: Cantharidin, cantharone 0.1%
  Arms: Part 1 Female; Part 1 Male

SUMMARY:
Inflammation is a key initiating and damaging factor in many illnesses including infection, arthritis and cancer but also of particular relevance to this study in diseases of the heart and blood vessels (i.e. cardiovascular disease). Much evidence now exists demonstrating that male sex increases ones risk of cardiovascular disease. More recent evidence demonstrates that inflammatory responses in females appear to dampened in comparison to age matched males. Since inflammation is thought to be a key initiating phenomenon in many cardiovascular disease states the investigators will examine the differences in acute inflammatory responses between the sexes in healthy volunteers and the impact this has on the function of blood vessels.

DETAILED DESCRIPTION:
We now know that one of the earliest events involved in precipitating disease of the heart and blood vessels is the phenomenon of inflammation and that this inflammation is a key process involved in dampening the protective nature of the inner lining (the endothelium) of the blood vessel wall, called endothelial dysfunction. In healthy arteries the endothelium releases a number of factors that maintain the health of the blood vessel. These factors act to keep the blood vessel in an open and dilated state and prevent the furring up of the vessel by actively inhibiting the cell components of the blood from collecting at the endothelium and blocking the flow of blood through the artery. Recent research in animals has demonstrated that one of the key components of inflammation i.e. the attraction of white cells, is reduced in females compared to males and that this is due to a reduced expression of key proteins called 'adhesion molecules', an in particular a molecule called P-selectin, on the endothelium. We now wish to determine whether similar differences in white cell attraction and adhesion molecules exist between the sexes in humans and whether these differences might underlie differences in endothelial function.

To investigate this possibility we will conduct a study in two parts, using well validated models of acute inflammation in healthy volunteers.

Part 1 To determine whether responses to inflammation differ between sexes in part 1 we will use a cantharidin-induced model of acute inflammation. Previous published studies have shown when cantharidin is applied to the skin it causes acantholysis and blister formation. It is a safe, reproducible technique with no permanent scarring or ill-effects. We will study the effects on inflammatory responses by measuring the levels of cells and inflammatory mediators in blister fluids, urine and plasma. Participants will given two blisters that will be harvested at 24 hours (acute phase) and 72 hours (resolution phase) after cantharidin application. The effects of inflammation on blood vessels will also be studied through non invasive blood pressure measurements.

Part 2 To determine whether susceptibility to inflammation-induced endothelial dysfunction is distinct between the sexes in part 2 we will use typhoid vaccine to induce mild inflammation throughout the body including the blood vessels. Previous published studies have shown that vaccination induces an acute inflammation that results in a temporary (reversed within 48h) dysfunction of the endothelium that can be measured using a range of non-invasive techniques called ultrasound flow-mediated dilatation and pulse wave velocity. We will use these techniques together with biochemical measurements to determine possible associations of endothelial dysfunction with specific inflammatory factors. In particular we will investigate the possibility that differences in the expression of the adhesion molecule P-selectin might have a role to play in differences between the sexes.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects aged 18-45 who have volunteered themselves and are willing to sign the consent form.

Exclusion Criteria:

1. Healthy subjects unwilling to consent
2. History of hypertension, diabetes or hypertensive on BP measurement
3. Pregnant, or any possibility that a subject may be pregnant unless in the latter case a pregnancy test is performed with a negative result
4. History of any serious illnesses, including recent infections or trauma
5. Subjects taking systemic medication (other than the oral contraceptive pill)
6. Subjects with self-reported use of mouthwash or tongue scrapes
7. Subjects with recent or current antibiotic use
8. Subjects with a history, or recent treatment of (within last 3 months) of any oral condition (excluding caries), including gingivitis, periodontitis and halitosis.
9. Subjects that have recently participated (preceding 3 months) in any clinical studies involving administration of an inflammogen.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Comparison change in blister fluid total and differential leukocyte numbers (Part 1) | 24, 72 h
  plasma and fluid collected from the blisters at 24 hours (acute phase) and 72 hours (resolution phase) after the cantharidin application will be analysed using standard laboratory techniques including flow cytometry
Flow-mediated dilatation (Part 2) | 0, 24, 48 h
  Flow mediated dilatation of the brachial artery will be assessed using ultrasound will be measured at time 0, 24 and 48h. At the 16h timepoint a single typhoid vaccination will be administered in the arm or buttock.

SECONDARY OUTCOMES:
Blood pressure (Part 1) | 0, 48, 72 h
  Blood pressure will be measured every 15 minutes for 1 hour
Platelet reactivity (Part 2) | 0, 24 and 48h
  Blood will be collected and platelet reactivity assessed using impedance aggreometry
Platelet activation (Part 2) | 0,24 and 48h
  Blood will be collected and platelet p-selectin and platelet-monocyte expression determined using flow cytometry
Arterial stiffness (Part 2) | 0, 24 and 48h
  The speed of blood pressure waves will be measured to give a pulse wave velocity measure for the aorta.
Inflammatory cell expression (Part 1 and 2) | 0, 48, 72h part 1, 0, 24 and 48h part 2
  Blood will be collected and inflammatory cell populations determined using flow cytometry
Blood inflammatory molecule expression (Part 1 and 2) | 0, 48, 72 h part 1, 0, 24 and 48h part 2,
  Plasma will be collected for assessment of inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, BSC PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- William Harvey Heart Centre, Barts & The London Medical School, London, United Kingdom

REFERENCES:
- [Background] Hingorani AD, Cross J, Kharbanda RK, Mullen MJ, Bhagat K, Taylor M, Donald AE, Palacios M, Griffin GE, Deanfield JE, MacAllister RJ, Vallance P. Acute systemic inflammation impairs endothelium-dependent dilatation in humans. Circulation. 2000 Aug 29;102(9):994-9. doi: 10.1161/01.cir.102.9.994. PMID 10961963
- [Derived] Rathod KS, Kapil V, Velmurugan S, Khambata RS, Siddique U, Khan S, Van Eijl S, Gee LC, Bansal J, Pitrola K, Shaw C, D'Acquisto F, Colas RA, Marelli-Berg F, Dalli J, Ahluwalia A. Accelerated resolution of inflammation underlies sex differences in inflammatory responses in humans. J Clin Invest. 2017 Jan 3;127(1):169-182. doi: 10.1172/JCI89429. Epub 2016 Nov 28. PMID 27893465